CLINICAL TRIAL: NCT05703009
Title: A Double-Blind, Placebo-Controlled, Crossover Study of Sacrosidase for the Treatment of Subjects With Fructan Intolerance
Brief Title: Effects of Sacrosidase and Placebo in Subjects With Fructan Intolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: QOL Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSDXA-14
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Fructan Intolerance
MeSH Terms: interventions — beta-Fructofuranosidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Subjects will be randomized to take active treatment, sacrosidase, 2 mL (17,000 IU) with every meal or snack, administered orally following dilution with 2 to 4 ounces (60 to 120 mL) of water or milk (either cold or at room temperature) during either Treatment Period 1 or Treatment Period 2. The study treatment period is one week.
  Interventions: Drug: Sacrosidase Oral Solution
- Placebo (Placebo Comparator): Subjects will be randomized to take placebo treatment, sacrosidase placebo, 2 mL (17,000 IU) with every meal or snack, administered orally following dilution with 2 to 4 ounces (60 to 120 mL) of water or milk (either cold or at room temperature) during either Treatment Period 1 or Treatment Period 2. The study treatment period is one week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sacrosidase Oral Solution — Study drug
  Other Names: sacrosidase
  Arms: Treatment
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
SSDXA-14 is a Phase 2 (feasibility/pilot) double-blind, placebo-controlled, crossover study to evaluate the efficacy and safety of sacrosidase and placebo in 25 subjects objectively diagnosed with fructan intolerance.

DETAILED DESCRIPTION:
This Phase 2 study will evaluate the efficacy and safety of sacrosidase and placebo in male and female subjects aged 18 years or older objectively diagnosed with fructan intolerance via fructan breath test within 6 months prior to informed consent and are negative for inflammatory bowel disease or low-grade GI bacterial infection, detected by fecal calprotectin test, celiac disease, detected by serology for anti-gluten protein antibodies, congenital sucrase-isomaltase deficiency (CSID), detected by sucrose hydrogen-methane breath test, and have a negative result for abnormal uncontrolled thyroid function, detected by the standard TSH blood test. This study will consist of a Screening Visit, Baseline Period, Treatment Period 1, Washout Period, and Treatment Period 2. Subjects will be required to attend 5 clinic visits during study participation. Subjects will be randomized in a 1:1 fashion to either receive sacrosidase or placebo during Treatment Period 1. Following a 7-day Washout Period, subjects will receive their crossover study medication for Treatment Period 2. Subjects will take their assigned study medication for 7 days during each Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and provide a signed and dated informed consent form
* Stated willingness to comply with all study procedures and attend all scheduled clinic visits, and continue participation for the duration of the study
* Ability to self-administer oral medication and willingness to adhere to the medication regimen
* Male or non-pregnant, non-lactating female, at least 18 years of age
* Sexually active women of childbearing potential must agree to use at least one reliable method of birth control while participating in the study
* Presence of fructan intolerance as determined by a positive result on a FBT within the last 6 months
* Subjects who are lactose intolerant agree to eliminate all lactose from their diet during the study
* Stated willingness to discontinue any medications to resolve GI symptoms (digestive enzymes, antacids, proton pump inhibitors, histamine-2 blockers, promotility agents, or anti-diarrheal agents, etc.), per the investigator's discretion.
* Stated willingness to discontinue any over the counter or prescribed oral nonsteroidal anti-inflammatory drugs (NSAIDs) during the study
* Per the discretion of the investigator, absence of any GI disorder other than a diagnosis of fructan intolerance

Exclusion Criteria:

* History of inflammatory bowel disease or active low-grade GI bacterial infection, as diagnosed by the presence of fecal calprotectin
* History of celiac disease, as diagnosed by serology testing for anti-gluten protein antibodies
* History of CSID, as diagnosed by the sucrose hydrogen-methane breath test,
* Abnormal uncontrolled thyroid function, detected by abnormal TSH level in the blood
* Per the discretion of the investigator, history of a serious physical or mental disorder
* BMI greater than 30 kg/m2
* History of diabetes
* History of hypersensitivity to yeast, yeast products, glycerin (glycerol), or papain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Change in incidence and severity of gastrointestinal symptoms in subjects with fructan intolerance treated with sacrosidase and placebo | Up to 7 weeks
  Change from baseline as determined by the Daily Symptom Questionnaire Total Symptom Score (TSS) rating severity on a scale from 0 to 9 and frequency on a scale from 0 to 5, based on a mean value of combination scores for, incidence of seven GI symptoms experienced in the past 24 hours during a 7-day period and severity of seven GI symptoms experienced in the past 24 hours during a 7-day period.

SECONDARY OUTCOMES:
Change in incidence and severity of abdominal pain in subjects with fructan intolerance treated with sacrosidase and placebo | Up to 7 weeks
  Change from baseline as determined by the Daily Symptom Questionnaire Total Symptom Score (TSS) rating severity on a scale from 0 to 9 and frequency on a scale from 0 to 5, based on a mean value of combination scores for, incidence of abdominal pain experienced in the past 24 hours during a 7-day period and severity of abdominal pain experienced in the past 24 hours during a 7-day period.
Assess the safety and tolerability of sacrosidase compared to placebo in subjects with fructan intolerance | Up to 1 year
  Frequency and severity of treatment emergent adverse events (TEAEs) and Serious Adverse Events (SAEs) and any premature study withdrawals related to adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Weng Tao, M.D., Ph. D, Principal Investigator — QOL Medical, LLC
Locations (1):
- Boston Specialists, Boston, Massachusetts, United States